CLINICAL TRIAL: NCT01448148
Title: Measuring the Impact of Cognitive and Psychosocial Interventions in Persons With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Laval University (Other)
Responsible Party: Principal Investigator, Sylvie Belleville, Research director of CRIUGM and full professor at University of Montreal, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRIUGM-002
Record Dates: First submitted 2011-09-28; First posted 2011-10-07 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive intervention (Experimental): Use of Memo protocol for 8 weeks
  Interventions: Other: Cognitive intervention
- Psychosocial intervention (Experimental): Use of "Programme d'intervention psychosociale axé sur le bien-être psychologique" for 8 weeks
  Interventions: Other: Psychosocial intervention
- no contact control group (No Intervention): waiting list

INTERVENTIONS:
Other: Cognitive intervention — Different strategies will be included to improve episodic memory. Training on imagery will be provided prior to episodic training.Particular attention will be paid to memory self-efficacy and the negative perception that elderly individuals entertain about memory tasks. The issue of generalization is of major importance in cognitive therapy.
  Arms: Cognitive intervention
Other: Psychosocial intervention — Based on a cognitive-behavioural approach, the psychosocial intervention will aim at improving general psychological well-being or preventing psychological distress in persons with MCI.
  Arms: Psychosocial intervention

SUMMARY:
Memory interventions are training programs that provide a variety of cognitive and psychological strategies meant to improve memory. These interventions have been shown to yield significant benefits to normal aged persons and small-size studies have shown that they are suitable and beneficial for persons with mild cognitive impairment. The goal of this proposal is to assess with a well-controlled design the efficiency and specificity of cognitive training in persons with mild cognitive impairment.

The hypothesis is that cognitive training can improve the cognition of persons with mild cognitive impairment and that this improvement can be enduring.

DETAILED DESCRIPTION:
Elderly persons with mild cognitive impairment experience a cognitive decline that is confirmed by a neuropsychological examination but do not meet the clinical criteria for dementia. However, longitudinal studies have shown that up to 75% of these persons develop dementia of the Alzheimer type after 5 years of follow-up. A significant proportion of these persons are thus in a prodromal phase of the disease. This phase is likely to represent a key moment in which to apply appropriate interventions. Indeed, these persons have the cognitive capabilities to benefit from such interventions. Cognitive training has been shown to be effective in improving the memory function of older persons without cognitive decline and increasing evidence indicates that persons with MCI might also benefit from such interventions. However, there is few researches have focused on the Mild Cognitive Impairment population in spite of the fact that they are at-risk of experiencing significant cognitive problems in the next few years while still having the potential to benefit from non-pharmacological interventions. In a number of pilot studies, the investigators compared cognitive and psychosocial intervention to a control intervention in persons with MCI. The participants' performance improved on proximal outcomes and on distal outcomes (activities of daily living). The purpose of this project is to study the efficacy of the cognitive intervention in a larger group of participants, compare it with a non-cognitive intervention, assess the long term maintenance of the improvement and measure the potential implication of cognitive and psychosocial factors.

Persons with Mild Cognitive Impairment will first receive a comprehensive clinical assessment to determine whether they meet the research criteria for Mild Cognitive Impairment. They will then be randomly allocated to one of three groups. One group will receive cognitive training, one group will receive psychosocial intervention and one group will receive no intervention. The two interventions will be offered on a one-session per week basis during an 8-week period. The cognitive intervention will include training of attention and episodic memory. This intervention is based on recently acquired knowledge regarding the nature of the deficits in mild cognitive impairment as well as factors that are known to optimize memory. The psychosocial intervention will focus on goal management. Booster sessions will be offered to the intervention groups after 3 and 6 months. Each intervention will act as social contact control group for the other intervention. The third group will receive no intervention and will be used as a no-contact control group.

All groups will undergo one pre-intervention assessment (1-2 week before beginning of intervention), one post-intervention assessment (1-2 week after end of intervention) and additional assessments one week after before the booster sessions and nine month following end of training. This last assessment will measure long-term retention of training and will assess the degree of change in the clinical profile of patients.

ELIGIBILITY:
Inclusion Criteria:

* francophone
* MCI identified by a doctor
* normal corrected vision
* good hearing

Exclusion Criteria:

* history of neurological disorder
* major psychiatric illness
* alcoholism
* general anesthesia in the previous six months
* significant impairment of physical mobility

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in memory measures | one week before and after intervention, and three and six months later
  Unrelated word list learning and Face-name memory tests

SECONDARY OUTCOMES:
generalization of therapeutic gains to everyday life | one week before and after intervention, and three and six months later
  Self-Evaluation Complaints Questionnaire, Activities of Daily Living- Prevention Instrument questionnaire, Multifactorial Memory Questionnaire tests and participants will be asked to press a button to record each occasion when they use a strategy in their daily lives.
Change in psychological health measures | one week before and after intervention, and 3 and 6 months later
  geriatric anxiety inventory, griatric depression scale and general well-being schedule tests

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Belleville, Ph.D., Principal Investigator — Centre de recherche Institut universitaire de geriatrie de Montreal; Carol Hudon, Ph.D., Study Director — Laval University, Psychology department
Locations (2):
- Canada (2):
  - Centre de recherche de l'Institut universitaire de geriatrie de Montreal, Montreal, Quebec
  - Centre hospitalier Robert-Giffard, Québec, Quebec

REFERENCES:
- [Background] Belleville S, Gilbert B, Fontaine F, Gagnon L, Menard E, Gauthier S. Improvement of episodic memory in persons with mild cognitive impairment and healthy older adults: evidence from a cognitive intervention program. Dement Geriatr Cogn Disord. 2006;22(5-6):486-99. doi: 10.1159/000096316. Epub 2006 Oct 16. PMID 17050952
- [Background] Belleville S. Cognitive training for persons with mild cognitive impairment. Int Psychogeriatr. 2008 Feb;20(1):57-66. doi: 10.1017/S104161020700631X. Epub 2007 Oct 25. PMID 17958927